# RESEARCH SUBJECT INFORMATION AND ASSENT FORM Student Assent

**TITLE:** Facilitating Employment for Youth with Autism: A Replication Study of an Internship Model to Identify Evidence Baseed Practices

VCU IRB NO.: HM15031

This form may have some words that you do not know. Please ask someone to explain any words that you do not know. You may take home a copy of this form to think about and talk to your parents about before you decide if you want to be in this study.

### What is this study about?

The reason for this study is to test job training for young people like you in a high school or in a community job training program.

We have asked you to be in this study because you:

- 1. Have Autism Spectrum Disorder diagnosis
- 2. Attend a Henrico, Hanover, or Chesterfield County High School or a Southeastern Cooperative Educational Program (SECEP) High School Classroom
- 3. Are between the ages of 18 and 21.

# What will happen to me if I choose to be in this study?

In this study you will be asked to take part in an assessments before you start your last year in high school. We will collect your name, address, date of birth, and ask you questions about yourself and your experiences in high school and the community. We will use that information to understand your work skills, abilities, and support needs. Then, you will receive work training in one of two programs. The first job training program is in your school. The second job training program is a 9-month internship in a community business. Project staff will assign you to one of the two job training programs. You will not have a choice of the program to which you are assigned. Once you complete the program, you will graduate from high school. We will keep in touch with you for one year after you graduate. We will ask you questions about your job, how much money you make, and how many hours you work. We will also ask you about the supports you need to work.

If you decide to be in this research study, you will be asked to sign this form. Do not sign the form until you have all your questions answered, and understand what will happen to you.

### What might happen if I am in this study?

The following are examples of issues that you may come across that might bother you. You may experience scheduling changes in your training program. You may also experience stress from:

- other students
- Coworkers
- your boss

• customers in your job training program.

# What do I get if I am in this study?

You will get some money for your time when we interview you. Also, either program may help you get a paying job faster.

### Will you tell anyone what I say or do?

We will not tell anyone the answers you give or the things you do except for your parents/guardians, your teachers and other people who help you. If you tell us that someone is hurting you, or that you might hurt yourself or someone else, by law we have to report that to people or agencies that might help you.

If we talk about this study at meetings or in writing, we will never use your name unless your parent or guardians have said it is ok for us to tell your name.

# Do I have to be in this study?

You do not have to be in this study. If you choose to be in the study you may stop at any time. No one will blame you or disapprove if you drop out of the study. If you decide to not be in the study, you will return to your regular school.

### Questions

If you have questions about being in this study, you can talk to the following persons or you can have your parent or another adult call:

Carol M. Schall, PhD Virginia Autism Resource Center Virginia Commonwealth University Richmond, VA 23284-2020 (804)828-4523 cmschall@vcu.edu

Do not sign this form if you have any questions. Be sure someone answers your questions.

# Assent: I have read this form. I understand the information about this study. I am willing to be in this study. Student name printed Student signature Date Name of Person Conducting Informed Assent Discussion / Witness, printed

| 2 |
|---------------|
| $\overline{}$ |
| 2015 |
| Ñ |
| 7/20 |
| $\overline{}$ |
| 4 |
| $\overline{}$ |
| o |
| RB |
| $\simeq$ |
| _ |
| ರ |
| $\mathcal{C}$ |
| > |
| (I) |
| the |
| ţ |
| _ |
| ed by |
| $\overline{}$ |
| ွှ |
| Ψ |
| pproved |
| 2 |
| ppro |
| $\circ$ |

| Signature of Person Conducting Informed Assent Discussion / Witness | Date |
|---|---|
| Principal Investigator Signature (if different from above) | Date |
| Please check the statement that reflects your opinion about videotaped. | being photographed or |
| I consent to be photographed and/or videotaped durin | ng this study. |
| I <i>do not consent</i> to be photographed and/or videotap | ed during this study. |
| Participant name printed Participant sign | nature Date |
| Name of Person Conducting Informed Consent<br>Discussion / Witness (Printed) | - |
| Signature of Person Conducting Informed Consent Discussion / Witness | Date |
| Principal Investigator Signature (if different from above) | Date |